CLINICAL TRIAL: NCT06657989
Title: Optimal Intensity of Reactive Balance Training for Healthy Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Avril Mansfield, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-5665
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-10

CONDITIONS: Accidental Falls
Keywords: Postural balance; Aging; Biomechanics; Rehabilitation
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High intensity reactive balance training (Experimental): Participants will complete 5 1-hour training sessions over 11 days. During each training session, participants will complete 36 multi-directional (left-, right-, and forward-fall) perturbations. Participants assigned to high-intensity RBT will experience perturbations at 150% of the multi-step threshold; for example, for a multi-step threshold of 2 m/s^2 the high intensity perturbation will be 3 m/s^2.
  Interventions: Behavioral: Reactive balance training
- Moderate intensity reactive balance training (Active Comparator): Participants will complete 5 1-hour training sessions over 11 days. During each training session, participants will complete 36 multi-directional (left-, right-, and forward-fall) perturbations. Participants assigned to moderate-intensity RBT will experience perturbations at 100% of the multi-step threshold; for example, for a multi-step threshold of 2 m/s^2 the high intensity perturbation will be 2 m/s^2.
  Interventions: Behavioral: Reactive balance training
- Walking control group (Sham Comparator): Participants assigned to the walking control group will complete 36 trials of unperturbed walking in each training session.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Reactive balance training — Reactive balance training involves clients experiencing repeated balance perturbations so that they can practice and improve control of reactions to avoid falling after a loss of balance.
  Other Names: Perturbation-based balance training
  Arms: High intensity reactive balance training; Moderate intensity reactive balance training
Behavioral: Walking — Overground walking
  Arms: Walking control group

SUMMARY:
Falls in daily life are a serious risk for older adults. A new type of balance training, called reactive balance training (RBT) involves people losing balance many times so that they can practice fast balance reactions, like stepping reactions. Differences in training program features might explain differences in the results of previous RBT studies. Training intensity is the difficulty or challenge of the training program. It would be valuable to know if high-intensity RBT improves balance reactions quickly. The main goal of this study is to see if more intense RBT improves balance reactions faster than less intense RBT. The investigators will compare how quickly people improve balance reactions between high- and moderate-intensity RBT, and between RBT and a control program that does not include RBT. The investigators will also test if the improvements in balance reactions last after the training program is over. The secondary goals are to understand exactly how balance reactions improve with training, and to determine if people who complete RBT improve their general balance skills, and falls efficacy more than people who do not complete RBT.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults (65-80 years old)

Exclusion Criteria:

* Unable to stand independently without upper-limb support for >30 seconds and/or walk independently (without a gait aid) for ≥10 metres;
* Diagnosed neurological condition that could affect balance control (e.g., stroke, Parkinson's disease);
* Score below normative values on the Montreal Cognitive Assessment;
* Score below age-matched normative values for sensory and motor function, as assessed using the FallScreen battery;
* Have insufficient English language comprehension such that they cannot understand instructions;
* Have contraindications to reactive balance training such as severe osteoporosis; and/or
* Are currently attending physiotherapy or supervised exercise.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of reactive steps | Two weeks
  Learning rate for number of steps to recover from 'backward fall' balance perturbations

SECONDARY OUTCOMES:
Step initiation time | One week and 12 weeks post-training
  Time from perturbation onset time to foot off time
Step execution time | One week and 12 weeks post-training
  Time from foot off to foot contact of the first step
Step length | One week and 12 weeks post-training
  Difference in foot position from foot off to foot contact
Braking impulse | One week and 12 weeks post-training
  Antero-posterior shear force generated over time on step contact
Mechanical margin of stability | One week and 12 weeks post-training
  Distance between the extrapolated centre of mass (incorporating centre of mass position and velocity) and the edge of the base of support
Balance evaluation systems test | One week and 12 weeks post-training
  Scale ranges from 0-100, with higher scores indicating better outcome
Falls efficacy scale - International | One week, 12 weeks, and 12 months post-training
  Scale range: 10-100; higher values indicate worse outcome

OTHER OUTCOMES:
Fall incidence | 12 months post-training
  Falls in daily life
Injurious fall incidence | 12-months post-training
5-level EuroQoL health status measure (EQ-5D-5L) | One week, 12 weeks, and 12 months post-training
  Scale range for descriptive component: 5-25, higher values indicate worse outcome; Scale range for visual analogue scale: 0-100, higher values indicate better outcome
Number of participants with fear of falling | One week, 12 weeks, and 12 months post-training
Number of participants with activity curtailment due to fear of falling | One week, 12 weeks, and 12 months post-training

CONTACTS AND LOCATIONS:
Overall Officials: Avril Mansfield, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No